CLINICAL TRIAL: NCT05487859
Title: A Pilot Study of the Immunomodulatory Agent Acarbose in Combination with Standard Therapy in Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Acarbose in Combination with Standard Therapy in Metastatic Renal Cell Carcinoma (RCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Arnab Basu, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB23143
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Ipilimumab (1 mg/kg) IV q3wks + Nivolumab (3mg/kg) IV q3wks + Acarbose (upto 100 mg PO TID) followed by Nivolumab 480 mg IV q4 wks + Acarbose (upto 100 mg PO TID)
  OR
  Pembrolizumab 200 mg IV q3 wks or 400 mg IV q6 wks + Lenvatinib (up to 20 mg PO Daily) + Acarbose (upto 100 mg PO TID) [ Frontline/Refractory pts]
  OR
  Lenvatinib (upto 18 mg PO daily) + Everolimus (upto 5 mg PO Daily) + Acarbose (upto 100 mg PO TID) [ Refractory pts]
  OR
  Cabozantinib (upto 60 mg PO Daily) + Acarbose (upto 100 mg PO TID) [Refractory pts]
  Interventions: Drug: Acarbose Tablets

INTERVENTIONS:
Drug: Acarbose Tablets — Acarbose Tablets PO ranging from 25 mg initially to 100 mg as tolerated

SUMMARY:
The purpose of this study is to determine the safety and tolerability of acarbose in combination of immunotherapy based standard of care therapy in advanced renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of clear cell or non-clear cell carcinoma of the kidney, except for medullary carcinoma, collecting duct carcinoma, lymphoma and sarcoma. Sarcomatoid features of any degree are allowed
2. Must have locally advanced or unresectable metastatic disease (i.e., newly diagnosed Stage IV RCC per American Joint Committee on Cancer) or has recurrent disease.
3. Has measurable disease per RECIST 1.1 as assessed by the investigator/site radiologist.
4. Has received no prior systemic therapy for advanced RCC in the past 3 weeks.
5. Has Karnofsky performance status (KPS) ≥ 60% as assessed within 10 days prior to randomization.
6. If receiving bone resorptive therapy (including but not limited to bisphosphonate or RANK-L inhibitor) must have therapy initiated at least 2 weeks prior to randomization.
7. Demonstrates adequate organ function defined as follows

   1. Liver function liver function (bilirubin < 3mg/dL, AST and/or ALT <3 x ULN)
   2. Kidney function (CrCL >=15ml/min using cockroft-gault method)
   3. ANC >= 500/microliter, Hemoglobin > 8 mg/dL, platelet count > 50,000/microliter
8. CNS metastasis is allowed if has been treated >3 weeks and patient has achieved clinical stability with no new neurologic deficits in the interim
9. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drugs. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* 1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization.

  2. Has had major surgery within 4 weeks, received radiation therapy within 2 weeks prior to randomization, or has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to prior treatment.

  3. Has a history of severe hypersensitivity reaction (e.g., generalized rash/erythema, hypotension, bronchospasm, angioedema or anaphylaxis) to acarbose or investigators choice of standard of care therapy.

  4. Has a diagnosis of immunodeficiency OR is receiving a systemic steroid therapy exceeding physiologic corticosteroid dose or any other form of immunosuppressive therapy within 7 days prior to randomization, except in the case of central nervous system (CNS) metastases.

  5. Has an active autoimmune disease requiring systemic treatment with in the past 2 years OR a documented history of clinically severe autoimmune disease. Note: Participants with vitiligo, Sjøgren's syndrome, Type 1 diabetes, resolved childhood asthma/atopy, hypothyroidism or adrenal or pituitary insufficiency who are stable on hormone replacement, are not excluded.

  6. Has a known additional malignancy that has progressed or has required active treatment in the last 3 years. Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer in situ are acceptable if they have undergone potentially curative therapy. Low grade prostate cancer with gleason score 6 or lower which is not under active therapy will be acceptable if in investigator judgement it is likely not a competing risk to patient's life expectancy.

  7. Has known active untreated CNS metastases and/or carcinomatous meningitis. 8. Has an active infection requiring systemic therapy. 9. Has received a live virus vaccine within 30 days of randomization. 10. Has a clinically significant gastrointestinal (GI) abnormality including Malabsorption, total gastric resection or any condition that might affect the absorption of orally taken medication.

  11. Active GI bleeding, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy 12. Has QT interval corrected for heart rate (QTc) ≥480 msec. 13. Has a history of any of the following cardiovascular conditions within 6 months of randomization: Myocardial infarction, Unstable angina pectoris Cardiac angioplasty or stenting, Coronary/peripheral artery bypass graft, Class III or IV congestive heart failure per New York Heart Association and Cerebrovascular accident or transient ischemic attack.

  14. Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥150 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg measured two times a day - despite the use of 3 or more antihypertensive medications.

  15. Has recorded hypoglycemic episodes with blood glucose <60 mg/dL documented within the last 12 months.

  16. Has medication treated diabetes and HbA1c < 8 gm/dL 17. Has hemoptysis within 6 weeks prior to randomization. 18. Has current use (within 7 days of randomization) or anticipated need for treatment with drugs or foods that are known strong cytochrome P450 (CYP3A4/5) inhibitors.

  19. Has current use (within 7 days of randomization) or anticipated need for treatment with drugs that are known strong CYP3A4/5 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort; or drugs that are known with proarrhythmic potential.

  20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

  21. Has had a prior solid organ transplant. 22. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety profile of acarbose in addition to standard of care (SOC) treatment in RCC | 2 years
  adverse events will be defined and assessed using the National Cancer Institute's Common Terminology Criteria (CTCAE) v5.0
To assess the effect of acarbose on the gut microbiome in patients receiving as standard of care therapy. | 2 years
  Fecal microbiota populations will be characterized prior, during and after treatment with acarbose.

SECONDARY OUTCOMES:
To assess the efficacy of Acarbose in combination with SOC treatment in RCC | 2 years
  Estimate of the median progression free survival (mPFS) of patients treated with SOC + Acarbose
To assess the efficacy of Acarbose in combination with SOC treatment in RCC | 2 years
  Estimate of the median overall survival (mOS) of patients treated with SOC + Acarbose

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No